CLINICAL TRIAL: NCT05299281
Title: Micropulse Transscleral Diode Laser Cyclophotocoagulation (MP-TSCPC) as a Treatment Modality for Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Gehad Hassan Abdelhalim Mohamed Youssef, Assisstant lecturer of ophthalmology, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS 9-222
Record Dates: First submitted 2022-03-09; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Glaucoma
Keywords: glaucoma; micropulse laser
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glaucoma patients (Other): Patients were enrolled from outpatient clinic with glaucoma during the period between January 2020 and July 2021
  Interventions: Device: Micropulse transscleral cyclophotocoagulation (MP-TSCPC)

INTERVENTIONS:
Device: Micropulse transscleral cyclophotocoagulation (MP-TSCPC) — patients undergone micropulse laser transscleral cyclophotocoagulation. The laser settings ranged from 2000- 2500 mW of 810 nm infrared diode laser radiation set on micro- pulse mode (Iris Medical Instruments, Mountain View, CA, USA), delivered over 100-200 s (envelope of micropulses) depending on severity of the case and other patient factors.
  Follow-up was done at day 1, week 1, month 1, month 3, and month 6 postoperatively.

SUMMARY:
The study objective was to evaluate the efﬁcacy and safety of transscleral cyclophotocoagulation (TSCPC) using micropulse diode laser treatment in patients with various types of glaucoma.

DETAILED DESCRIPTION:
Evaluation of the efﬁcacy and safety of a new form of transscleral cyclophotocoagulation (TSCPC) using micropulse diode laser treatment in patients with various types of glaucoma.

In this study, 810 nm infrared diode laser radiation in the micro- pulse mode was used in conjunction with a G probe (IRIDEX Medical Instruments, Mountain View, CA, USA).

The laser settings ranged from 2000- 2500 mW of 810 nm infrared diode laser set on micro- pulse mode, delivered over 100-200 seconds (envelope of micropulses) depending on severity of the case and other patient factors. With duty cycle 31.3% (This translates to 0.5 ms "on" time and 1.1 ms "off" time), which allows the tissue to cool down between laser shots, thus greatly reducing thermal damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with glaucoma if they had uncontrolled Intraocular pressure despite maximal tolerated medical therapy.
* Patients who are unable to maintain compliance with the prescribed topical medications.
* Patients who need filtering glaucoma surgery for controlling Intraocular pressure but are not generally fit for the surgery.
* Patients who refused incisional procedures like subscleral trabeculectomy.

Exclusion Criteria:

* Patients who were unable to give informed consent.
* Patients who had undergone previous conventional transscleral diode laser cyclophotocoagulation (TSCPC).
* Patients with signiﬁcant scleral thinning deﬁned as thinning of more than one clock hour noticed on scleral transillumination.
* Patients with ongoing ocular infection or inflammation.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | Follow-up was done at day 1, week 1, month 1, month 3, and month 6 postoperatively
  significant change in IOP in mmHg.
best corrected visual acuity (BCVA) | Follow-up was done at day 1, week 1, month 1, month 3, and month 6 postoperatively
  change in BCVA using snellen's chart

SECONDARY OUTCOMES:
complication rate. | Follow-up was done at day 1, week 1, month 1, month 3, and month 6 postoperatively
  Describing any complications related to the procedure.
change in number of postoperative glaucoma medications. | Follow-up was done at day 1, week 1, month 1, month 3, and month 6 postoperatively
  Number of postoperative glaucoma medications.
retreatment rate. | Follow-up was done at day 1, week 1, month 1, month 3, and month 6 postoperatively
  percentage of patients needing further treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gehad H Youssef, Msc, Principal Investigator — Benha University
Locations (1):
- Benha University, Banhā, Other, Egypt

IPD SHARING:
Plan to Share IPD: No